CLINICAL TRIAL: NCT07298291
Title: A Phase 1, Single-Center, Prospective Study to Evaluate the Safety and Clinical Utility of Anterior Chamber Paracentesis for Proteomic Analysis in Patients With Geographic Atrophy Secondary to Dry Age-Related Macular Degeneration
Brief Title: Ocular Proteomics Testing In Chronic Atrophy
Acronym: OPTICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ClinOmicsAI (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: COAI-OPTICA-001
Record Dates: First submitted 2025-12-01; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Age-Related (Dry) Macular Degeneration
Keywords: geographic atrophy; AMD
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GA patients (Experimental): Anterior chamber paracentesis (ACP)
  Interventions: Procedure: AC Tap (anterior chamber paracenthesis)

INTERVENTIONS:
Procedure: AC Tap (anterior chamber paracenthesis) — anterior chamber paracenthesis (microvolume of eye fluid is taken)

SUMMARY:
Study to evaluate the safety of routine diagnostic anterior chamber paracentesis (ACP) for proteomic profiling in patients with geographic atrophy (GA)

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and tolerability of serial (two) AC paracentesis procedures, performed at Baseline and Month 1, for the collection of AH in subjects with Geographic Atrophy (GA) or dry Age-Related Macular Degeneration (dAMD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 50 and 89 years, inclusive
* For the GA cohort: Clinical diagnosis of GA secondary to AMD or dAMD in the study eye, confirmed by fundus autofluorescence imaging and spectral-domain optical coherence tomography (SD-OCT).
* For the control cohort: No clinical evidence of retinal disease in either eye.
* Best-corrected visual acuity (BCVA) of ≥20/200 in the study eye, as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) charts
* Ability and willingness to provide written informed consent before any study-specific procedures.

Exclusion Criteria:

* Presence of active ocular infection or inflammation in either eye at the time of screening.
* History of intraocular surgery in the study eye within the three months preceding enrollment.
* Intraocular pressure (IOP) greater than 21 mmHg in the study eye at screening
* Use of systemic anticoagulation therapy that cannot be safely discontinued prior to ACP.
* Pregnant or nursing women.
* Known hypersensitivity or contraindication to any of the medications or procedures used in the study.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From enrollment to end of Visit 2
  Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Longitudinal changes in the Aqueous Humor proteome between Baseline (Day 0) and Month 1 (Day 30) | From Baseline (Day 0) to Month 1 (Day 30)
  The secondary objective of this study is to characterize longitudinal changes in the AH proteome between Baseline (Day 0) and Month 1 (Day 30) by analyzing AH specimens collected at these two time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Erie Retina Research, Erie, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Exploratory study only